CLINICAL TRIAL: NCT06589635
Title: A Single-center, Open-label and Sequential-dosing Clinical Trial Investigating the Drug Interaction Between ADC-189 Tablet and Itraconazole Capsule in Healthy Adult Subjects
Brief Title: A Drug-Drug Interaction (DDI) Study of ADC189 With Itraconazole in Healthy, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiaxing AnDiCon Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-ADC189-I-002
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-06

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ADC-189 and itraconazole (Experimental): Part 1: Single dose of ADC-189
  Part 2: Itraconazole with single dose of ADC-189
  Interventions: Drug: ADC-189 and Itraconazole

INTERVENTIONS:
Drug: ADC-189 and Itraconazole — Part 1:
  Day 1, fasting condition, 45 mg ADC189, administered orally
  Part 2:
  Day 22, 200 mg itraconazole bid, taken orally after meals. Day 23-Day 25, 200 mg itraconazole was taken orally after meals. Day 26, 45 mg ADC-189 and 200 mg itraconazole was taken orally after meals. Day 27-Day 39, 200 mg itraconazole was taken orally after meals.
  Other Names: Part 1: Single dose of ADC-189; Part 2: Itraconazole with single dose of ADC-189

SUMMARY:
This study aims to answer how repeat doses of itraconazole impact the pharmacokinetics, safety, and tolerability of single doses of ADC189 in healthy adults.

Participants in this study will complete screening assessments within 14 days before the first dose of ADC189. Participants will be admitted to the clinical pharmacology center (CPC) and complete 2 periods of treatments. On Day 1 and 26, each participant will receive a single oral dose of ADC189 (45mg), under fasting condition On Day 22, all participants will receive oral doses of itraconazole 200 mg (bid), after meal. From Day 23 to Day 25, and Day 26-D39, participants will receive itraconazole 200 mg(qd). Blood and safety assessments will continue for 336-hours after dosing on Day 1 and Day 26. Participants will receive a telephone follow-up on D47 (±3) days for a final visit.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent, be capable of and willing to comply with study restrictions and procedures.
* Healthy adult subjects aged 18 to 55 years.
* Weight >=50kg for males, and >=45kg for females, BMI 19-26 kg/m^2.
* No clinical significance in physical examination, vital signs, laboratory examination, 12-lead electrocardiogram, abdominal ultrasound, and chest X-ray examination.

Exclusion Criteria:

* Subjects who participated in other drug trials within 3 months before screening
* Hospital admission or major surgery within 4 weeks prior to screening or a preplanned hospital admission during study participation
* Donated or lost ≥400 mL of blood in the previous 3 months before screening
* Have a history of allergic diseases (asthma, urticaria, eczema, etc.), or food allergies
* A history of drug abuse in the past five years
* Any condition or finding that in the Investigator's opinion would put the participant or study conduct at risk if the participant were to participate in the study
* Unable to complete this study for other reasons or the Investigator believes that he or she should be excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
AUC[0-∞] of ADC-189 | Part 1: Day 1 to Day 15; Part 2: Day 21 to Day 40
  Pharmacokinetics (PK) parameter: Area under the curve from time 0 hour to ∞
Cmax of ADC-189 | Part 1: Day 1 to Day 15; Part 2: Day 21 to Day 40
  PK parameter: Maximum observed concentration
AUC[0-t] of ADC-189 | Part 1: Day 1 to Day 15; Part 2: Day 21 to Day 40
  PK parameter: Area under the curve from time 0 to 336 hour
Adverse events (AEs) | Day 1 to Day 43
  Number of subjects reporting AEs

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affilicated Hospital of Bengbu Medical University
Locations (1):
- The First Affilicated Hospital of Bengbu Medical University, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No